CLINICAL TRIAL: NCT03853005
Title: Effect of High Volume Hemodiafiltration on Lung Oxygenation, Lung Mechanics and Biomarkers in Mechanically Ventilated Patients With Severe Sepsis
Brief Title: Effect of High volumeHemodiafiltration on Lung Oxygenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayman Abd El-Khalek Mohammed Glala, Ayman Abd ELkhalek Mohammed, lecturer, clinical anesthesiologist and principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 28503011700371A1
Record Dates: First submitted 2018-07-10; First posted 2019-02-25 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Haemofiltration; Lung Mechanics; Septic Patients
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (controlled group) (Placebo Comparator): They will not receive HVHDF treatment
  Interventions: Other: controlled
- Group B (HVHDF group) (Active Comparator): They will receive HVHDF treatment for 48 hours. HVHDF will be performed via indwelling central venous catheter. The blood flow will be 180-240 ml/min, and ultrafiltration rate will be 70 ml/kg/h during HVHF. The substitute fluid will be infused with pre-dilution. Heparin will be used for anti-coagulation, whose initial dose will be 15-25 U/kg, and maintenance dose is 5-15 U/kg/h. aPTT time maintained between 60-80 second and will be checked every 12 hours. The survival status of all of the subjects were followed up at 28 days after being diagnosed as severe sepsis.
  Interventions: Other: HVHDF

INTERVENTIONS:
Other: HVHDF — Patients will receive HVHDF treatment for 48 hours. HVHDF will be performed via indwelling central venous catheter. The blood flow will be 180-240 ml/min, and ultrafiltration rate will be 70 ml/kg/h during HVHF. The substitute fluid will be infused with pre-dilution. Heparin will be used for anti-coagulation, whose initial dose will be 15-25 U/kg, and maintenance dose is 5-15 U/kg/h. aPTT time maintained between 60-80 second and will be checked every 12 hours.
  Arms: Group B (HVHDF group)
Other: controlled — Patients will receive the usual care
  Arms: Group A (controlled group)

SUMMARY:
High volume hemodiafiltration (HVHDF) has been used in septic patients to get hemodynamic improvement and possibly survival benefit.

DETAILED DESCRIPTION:
Sepsis, defined as life-threatening organ dysfunction caused by dysregulated immune response to infection. Hemofiltration has been suggested as beneficial in restoring immune homeostasis. High volume hemodiafiltration (HVHDF) is a hybrid method of intermittent renal replacement therapy (RRT), where high filtration volumes are applied. In several studies; higher filtration volumes have been shown to achieve hemodynamic improvement and possibly survival benefit in patients with septic shock.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years
2. Severe sepsis defined by Quick SOFA score by presentation of 2 or more of the following criteria:

   * Mental clouding: decreased glasco coma scale GCS < 15
   * Hypotension: Systolic blood pressure < 100 mmgH
   * Tachypnea: respiratory rate > 22 breath/ minute Then serum lactate is analysed to confirm sepsis hypoperfusion if ≥ 2mmol/L
3. Organs dysfunction (including one of them respiratory failure).

Organ dysfunctions are defined as following:

Respiratory dysfunction (criteria for ARDS):

* PaO2/FiO2 <200
* Bilateral infiltrates in chest X-ray
* Resistant hypoxemia
* Tachypnoea (RR > 40 breath/minute)
* The need for invasive mechanical ventilation
* Excluded cardiac causes of pulmonary edema

CNS failure:

* Decreased GCS ≥ 4 decreased points

CVS dysfunction:

* Sustained hypotension even on very high inotropes doses (Noradrenaline >1µm/min)+ adrenaline>1.5µm/min associated
* with high CVP pressure > 12 mmHg and not responding to fluid challenge test to exclude hypovolemia.
* Cardiomegaly detected by either echocardiography assessment, or chest X-ray
* Resistant frequent ventricular ectopics not explained by organic causes.

Liver dysfunction:

* Elevated total and direct bilirubin than double normal or basal levels
* Elevated prothrombin time > 17 seconds or INR > 1.5
* Elevated liver enzymes > triple normal level

Renal dysfunction:

* Decreased urine output < 0.5 ml/kg.
* Elevated creatinine level > 164 µmol/L (1.5mg/dL).
* Decreased creatinine clearance <50ml/minute if available.

Bone marrow depression:

* Decreased platelets < 90 X 103/µL
* Decreased leukocytes <4 X 103/µL
* Decreased RBCs count < 4 X 106/µL

Exclusion Criteria:

1. Patient relatives' refusal
2. Pregnancy
3. Recent active internal hemorrhage
4. Not mechanically ventilated.
5. Hypersensitivity to the dialyser fluid

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
Arterial oxygen pressure (PaO2) | 24 hours after start of HVHDF
  Change in arterial oxygen pressure (PaO2) in units of millimeter mercury (mmHg)

SECONDARY OUTCOMES:
The ratio of arterial oxygen pressure to the fraction of inspired oxygen (PaO2/ FiO2 ratio) | 0 hour, 24 hours, and 48 hours after start of HVHDF
  Changes in the ratio of arterial oxygen pressure to the fraction of inspired oxygen (PaO2/ FiO2 ratio)
Ventilatory function | 0 hour, 24 hours, and 48 hours after start of HVHDF
  Changes in compliance (ml/cmH2O)
The duration for weaning from mechanical ventilation (MV) | 28 days
  Days until weaning the patient from mechanical ventilation (MV)

OTHER OUTCOMES:
Interleukin-6 | 0 hour, 24 hours, and 48 hours after start of HVHDF
  Changes in Interleukin-6 (ng/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Assiut university A Egypt, Study Director — Assiut University
Locations (1):
- Faculty of medicine - Assiut university, Asyut, Egypt